CLINICAL TRIAL: NCT04693065
Title: Pronostic Factors of Long Term Outcome in Patients With Clubfoot Treated by the Ponseti Method
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20_5080
Record Dates: First submitted 2020-09-18; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-09

CONDITIONS: Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ponseti: Patients treated by ponseti method
  Interventions: Other: ponseti

INTERVENTIONS:
Other: ponseti — Standard of care, treatment by ponseti method

SUMMARY:
We aim at finding prognostic factors of long term (after growth) function outcome in patient with clubfoot treated by ponseti method, based on a very complete prospective recording of treatment variables and outcome

ELIGIBILITY:
Inclusion Criteria:

* - Patients treated by ponseti method for clubfoot-

Exclusion Criteria:

* - other malformation associated / congenital

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by ponseti method
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Function at >16 years | at 18 years old or complete bone maturity
  Composite score (perfect or non-perfect function), perfect foot defined as a plantigrade, non painful, valgus barefoot with >10° dorsal flexion. Non-perfect otherwise.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital femme mere enfants, Lyon, France